CLINICAL TRIAL: NCT03461601
Title: The Impact of Uterine Flushing With Human Chorionic Gonadotrophin Before Intrauterine Insemination on Pregnancy and Live Birth Rates in Women With Unexplained Infertility: A Randomized Controlled Trial
Brief Title: Uterine Flushing With Human Chorionic Gonadotrophin and Unexplained Infertility
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ahmed Walid Anwar Murad (Other)
Responsible Party: Sponsor-Investigator, Ahmed Walid Anwar Murad, Assistant Professor, Department of Obstetrics and Gynecology, Faculty of Medicine; Banha University, Benha University
Organization: Benha University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 18144
Record Dates: First submitted 2018-02-28; First posted 2018-03-12 (Actual); Last update posted 2018-03-12 (Actual); Status verified 2018-03

CONDITIONS: Unexplained Infertility
MeSH Terms: interventions — Saline Solution

STUDY DESIGN:
Intervention Model Description: intrauterine injection of human chorionic gonadotropin before intrauterine insemination (IUI) compared to IUI alone
Who Masked: Participant
Masking Description: Vaginal flushing with 10 ml saline was performed in the control group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- HCG uterine flushing group (Active Comparator): Uterine flushing was done one day before Intrauterine insemination (IUI) with HCG (500 IU) in 10 ml of saline followed by Intrauterine insemination (IUI).
  Interventions: Procedure: HCG Uterine flushing; Procedure: IUI
- IUI alone group (Placebo Comparator): Intrauterine insemination alone plus vaginal flushing with 10 ml normal saline
  Interventions: Procedure: IUI; Procedure: Vaginal flushing with 10 ml normal saline

INTERVENTIONS:
Procedure: HCG Uterine flushing — HCG Uterine flushing was done one day before IUI with HCG (500 IU) in 10 ml of saline.
  Arms: HCG uterine flushing group
Procedure: IUI — Intrauterine insemination (IUI)
Procedure: Vaginal flushing with 10 ml normal saline — Flushing of the vagina with 10 ml of saline
  Arms: IUI alone group

SUMMARY:
A prospective randomized study included 210 women with Unexplained infertility subjected to combined ovarian stimulation and Intrauterine insemination (IUI). Two equal groups. Study group, subjected to uterine flushing with Human chorionic gonadotropin (HCG) one day before IUI and control group subjected to IUI alone.

DETAILED DESCRIPTION:
A prospective randomized study included 210 patients with Unexplained infertility subjected to coupled ovarian stimulation and Intrauterine insemination (IUI). Two equal groups. Study group, subjected to uterine flushing with Human chorionic gonadotropin (HCG) one day before IUI and control group subjected to IUI alone.

ELIGIBILITY:
Inclusion Criteria:

* Unexplained infertility (UI)

Exclusion Criteria:

* body mass index (BMI) ≥35 kg/m2,
* Follicle Stimulating Hormone >10 International Unit /Litter in early follicular phase,
* diagnosed cause of infertility, menstrual cycle irregularity,
* ovarian cysts,
* sever cervical stenosis,
* former IUI,
* ongoing pregnancy and
* renal or hepatic diseases were all the exclusion criteria.

Ages: 18 Years to 37 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 210 (Actual)
Dates: Start 2014-06-01 (Actual); Primary Completion 2017-06-01 (Actual); Study Completion 2017-06-01 (Actual)

PRIMARY OUTCOMES:
Live birth | 10 months of randomization
  Defined as pregnancies maintained beyond 20 weeks of gestation

SECONDARY OUTCOMES:
Chemical pregnancy | One month after randomization
  Defined as positive serum pregnancy test
Clinical pregnancy | Two months after randomization
  Defined by the presence of gestational sac with fetal heartbeats on ultrasound scan or histological identification of trophoblastic tissue.
Adverse effects | one hour of the procedure
  Nausea, vomiting, and pain